CLINICAL TRIAL: NCT01266265
Title: A Postmarketing Observational Study to Assess Respiratory Tract Adverse Events in Pulmonary Arterial Hypertension Patients Treated With Tyvaso® (Treprostinil) Inhalation Solution
Brief Title: Study of Incidence of Respiratory Tract AEs in Patients Treated With Tyvaso® Compared to Other FDA Approved PAH Therapies
Acronym: Aspire
Status: Completed | Type: Observational
Sponsor: United Therapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: RIN-PH-403
Record Dates: First submitted 2010-12-22; First posted 2010-12-24 (Estimated); Results first posted 2016-02-17 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2016-01

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: pulmonary arterial hypertension; PAH; treprostinil sodium; Tyvaso; inhalation; Ventavis; iloprost; prostacyclin; epoprostenol sodium; Flolan; Veletri; subcutaneous and intravenous prostacyclin analogue; Remodulin; oral ERA; bosentan; Tracleer; ambrisentan; Letairis; oral PDE5 inhibitors; sildenafil; Revatio; tadalafil; Adcirca; Opsumit; macitentan; Adempas; riociguat; Orenitram; oral treprostinil
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Respiratory Aspiration | interventions — treprostinil; Iloprost; Epoprostenol; Injections, Subcutaneous; Bosentan; ambrisentan; Phosphodiesterase 5 Inhibitors; Sildenafil Citrate; Tadalafil

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Tyvaso: The Tyvaso group will consist of patients receiving Tyvaso and may be receiving another FDA approved PAH therapy as part of routine care.
  Interventions: Drug: inhaled prostacyclin
- Control: The control group will consist of patients with no previous Tyvaso exposure and not taking Tyvaso at the time of the Baseline visit, but receiving any other FDA approved PAH therapy as part of routine care.
  Interventions: Drug: inhaled prostacyclin; Drug: prostacyclin; Drug: subcutaneous and intravenous prostacyclin; Drug: oral ERA; Drug: oral PDE5 inhibitors

INTERVENTIONS:
Drug: inhaled prostacyclin — Tyvaso
  Other Names: treprostinil
  Groups: Tyvaso
Drug: inhaled prostacyclin — As prescribed by the physician
  Other Names: iloprost, Ventavis
  Groups: Control
Drug: prostacyclin — As prescribed by the physician
  Other Names: epoprostenol sodium, Flolan
  Groups: Control
Drug: subcutaneous and intravenous prostacyclin — As prescribed by physician
  Other Names: treprostinil , Remodulin
  Groups: Control
Drug: oral ERA — As prescribed by physician
  Other Names: bosentan, Tracleer; ambrisentan, Letairis
  Groups: Control
Drug: oral PDE5 inhibitors — As prescribed by physician
  Other Names: sildenafil, Revatio; tadalafil, Adcirca
  Groups: Control

SUMMARY:
A surveillance of respiratory tract related adverse events in patients treated with Tyvaso®(treprostinil) Inhalation Solution versus other FDA approved therapies

DETAILED DESCRIPTION:
A post marketing surveillance to determine the type and incidence of oro/nasopharyngeal or pulmonary adverse events that may occur in patients treated with commercially available Tyvaso®(treprostinil) Inhalation Solution. A comparison will be made to the type and incidence of events in patients receiving other FDA approved therapies for pulmonary arterial hypertension, as a control measure.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of PAH, WHO GROUP I
* Prescribed and is currently receiving Tyvaso and/or other FDA-approved therapy for the treatment of PAH
* Willing and able to provide written informed consent

Exclusion Criteria:

* Previous initiation and permanent discontinuation of Tyvaso
* Participation in an investigational clinical drug or device trial within 30 days of enrollment
* Current or past diagnosis of lung neoplasm
* Active gastrointestinal or pulmonary bleed at enrollment
* Planned surgical intervention for treatment of PAH e.g., atrial septostomy or transplant

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: community centers, academic institutions
Sampling Method: Non-Probability Sample
Enrollment: 1333 (Actual)
Dates: Start 2010-12; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (88):
- United States (88):
  - Cardiovascular Associates, P.C., Birmingham, Alabama
  - The University of Alabama at Birmingham, Birmingham, Alabama
  - University of South Alabama, Mobile, Alabama
  - Arizona Pulmonary Specialists, LTD, Phoenix, Arizona
  - Berkeley Cardiovascular Medical Group, Berkeley, California
  - Cedars-Sinai Heart Institute, Beverly Hills, California
  - University California San Francisco, Fresno, California
  - University of Southern California, Los Angeles, California
  - West Los Angeles VA Healthcare Center, Los Angeles, California
  - University of California Davis Medical Center, Sacramento, California
  - University of California, San Francisco, San Francisco, California
  - Paloma Medical Group, San Juan Capistrano, California
  - Santa Barbara Cottage Hospital, Santa Barbara, California
  - Stanford Hospital and Clinics, Stanford, California
  - Children's Hospital Denver, Denver, Colorado
  - Western States Clinical Research, Inc., Wheat Ridge, Colorado
  - St. Francis Sleep Allergy & Lung, Clearwater, Florida
  - University of Florida, Gainesville, Florida
  - Pulmonary and Critical Care Associates, Jacksonville, Florida
  - University of Florida College of Medicine Jacksonville, Jacksonville, Florida
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Miami Center for Cardiovascular Disease, Miami, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Central Florida Pulmonary Group, P.A., Orlando, Florida
  - Orlando Heart Center, Orlando, Florida
  - Cleveland Clinic Florida, Weston, Florida
  - Emory University School of Medicine, Atlanta, Georgia
  - Georgia Lung Associates, PC, Austell, Georgia
  - Northwestern Medical Center, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Illinois at Chicago, Chicago, Illinois
  - Midwest Heart Foundation, Oakbrook Terrace, Illinois
  - Indiana University Hospital, Carmel, Indiana
  - University of Iowa, Iowa City, Iowa
  - Mercy Hospital, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Kentuckiana Pulmonary Associates, Louisville, Kentucky
  - University of Maryland, Baltimore, Maryland
  - Johns Hopkins University, Baltimore, Maryland
  - Tufts - New England Medical Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - William Beaumont Hospital, Troy, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Nebraska Pulmonary Specialties, LLC, Lincoln, Nebraska
  - Hackensack University Medical Center, Hackensack, New Jersey
  - UMDNJ - Robert Wood Johnson Medical Center Clinical Research Center, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - SUNY Stony Brook University Medical Center, Islandia, New York
  - Winthrop Pulmonary Associates, Mineola, New York
  - North Shore - Long Island Jewish Health System, New Hyde Park, New York
  - St. Luke's-Roosevelt Hospital Center, New York, New York
  - Columbia University Medical Center, New York, New York
  - Mary M Parkes Center, Rochester, New York
  - Pulmonary Health Physicians, Syracuse, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Pinehurst Medical Clinic, Pinehurst, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Akron General Hospital, Akron, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Davis Heart and Lung Research Institute, Columbus, Ohio
  - Mercy Fairfield Hospital, Fairfield, Ohio
  - Legacy Pulmonary Northwest, Portland, Oregon
  - Oregon Clinic, PC, Portland, Oregon
  - OHSU-Oregon Health and Science University, Portland, Oregon
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Pennsylvania Health System, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Temple University, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Berks Schuylkill Respiratory Specialists, Ltd., Wyomissing, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Lexington Pulmonary and Critical Care, Lexington, South Carolina
  - MD Total Care, PLLC, Chattanooga, Tennessee
  - Summit Medical Group, Knoxville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - UT Southwestern Medical Center, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - Texas Children's Hospital, Houston, Texas
  - University of Texas Health Science Center at Houston, Houston, Texas
  - Methodist Healthcare System of San Antonio, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Sentara Cardiovascular Research Institute, Norfolk, Virginia
  - Aurora Health Care, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Zamanian RT, Levine DJ, Bourge RC, De Souza SA, Rosenzweig EB, Alnuaimat H, Burger C, Mathai SC, Leedom N, DeAngelis K, Lim A, De Marco T. An observational study of inhaled-treprostinil respiratory-related safety in patients with pulmonary arterial hypertension. Pulm Circ. 2016 Sep;6(3):329-37. doi: 10.1086/688059. PMID 27683610

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period for this study was February 2010 to December 2014. All sites were located in the United States.
Groups:
- Control: The control group will consist of patients with no previous Tyvaso exposure and not taking Tyvaso at the time of Baseline visit, but treated with any other FDA approved PAH therapy as part of routine care.
  inhaled prostacyclin: As prescribed by the physician prostacyclin: As prescribed by the physician subcutaneous and intravenous prostacyclin: As prescribed by physician oral ERA: As prescribed by physician oral PDE5 inhibitors: As prescribed by physician
Period: Overall Study
Arm/Group | Tyvaso | Control
Started | 666 | 667
Completed | 461 | 477
Not Completed | 205 | 190
Not completed — Death | 95 | 73
Not completed — Lost to Follow-up | 23 | 28
Not completed — Withdrawal by Subject | 13 | 11
Not completed — Respiratory-related adverse event | 2 | 1
Not completed — Transferred care to another provider | 22 | 28
Not completed — Stopped/changed PAH medication(s) | 16 | 9
Not completed — Enrolled in another clinical study | 15 | 26
Not completed — Non-compliance | 8 | 5
Not completed — Lung transplant | 6 | 5
Not completed — Site closed early | 4 | 3
Not completed — Clinical worsening | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tyvaso | Control | Total
Number analyzed (Participants) | 666 | 667 | 1333
Age, Continuous [Median (Full Range); unit: years] | 57.5 [5 to 90] | 57.0 [3 to 97] | 57.25 [3 to 97]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 519 | 532 | 1051
  Male | 147 | 135 | 282
Disease etiology [Number; unit: participants] — Patients were instructed to select all that apply.
  participants
    Idiopathic/heritable/drug- or toxin-induced | 341 | 389 | 730
    Connective tissue disease | 223 | 195 | 418
    Congential heart disease | 55 | 37 | 92
    HIV infection/porto-pulmonary | 53 | 55 | 108
    Other | 9 | 4 | 13
Race [Number; unit: participants] — Patients were instructed to select all that apply.
  participants
    White | 483 | 510 | 993
    Black/African American | 116 | 107 | 223
    Other/race not disclosed | 42 | 33 | 75
    Asian | 21 | 15 | 36
    Native Hawaiian/Pacific Islander | 3 | 1 | 4
    American Indian/Alaska Native | 2 | 1 | 3
Years Since PAH Diagnosis [Median (Full Range); unit: years] | 2.9 [0 to 32.0] | 2.9 [0 to 26.0] | 2.9 [0 to 32.0]
Baseline PAH Medication [Number; unit: participants] — Patients were instructed to select all that apply.
  participants
    Tyvaso (treprostinil) inhalation | 666 | 0 | 666
    Remodulin (treprostinil) | 2 | 150 | 152
    Flolan (epoprostenol) | 2 | 44 | 46
    Veletri (epoprostinol) | 0 | 36 | 36
    Ventavis (iloprost) inhalation | 0 | 33 | 33
    Revatio (sildenafil citrate) | 294 | 236 | 530
    Adcirca (tadalafil) | 239 | 224 | 463
    Letairis (ambrisentan) | 250 | 200 | 450
    Tracleer (bosentan) | 164 | 203 | 367
    Opsumit (macitentan) | 4 | 2 | 6
    Adempas (riociguat) | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Prevalence of Respiratory Tract-Related Adverse Events of Interest
Description: Percentage of patients who experienced a respiratory tract-related adverse event (grouped by category of interest) during the study.
Time Frame: Follow-up every 3 months
Measure: Number; unit: percentage of participants
Arm/Group | Tyvaso | Control
Number analyzed (Participants) | 666 | 667
percentage of participants
  Any Event | 52 | 51
  Bleeding from the upper or lower respiratory tract | 16 | 14
  Irritation/pain of nose, mouth, larynx, pharynx | 17 | 10
  Upper or lower respiratory tract infection | 37 | 40
  Wheezing, bronchospasm, or asthma/COPD exacerbate | 12 | 13

ADVERSE EVENTS:
Time Frame: Respiratory tract-related AEs were recorded from the time of informed consent to study completion or discontinuation.
Description: SAEs were included in the "Other" AE table because one participant may have experienced both an SAE and non-serious AE during the study. Non-respiratory-related AEs and SAEs were outside the scope of this study.
Arm/Group | Tyvaso | Control
Serious Adverse Events (participants affected / at risk) | 96/666 | 94/667
Other Adverse Events (participants affected / at risk) | 403/666 | 388/667
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tyvaso (N=666) | Control (N=667)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 42 (45) | 37 (45)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 13 (18) | 7 (9)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 12 (13) | 10 (10)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 9 (12) | 7 (10)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 (10) | 8 (12)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 3 (3)
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 6 (6)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 5 (5)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 5 (5)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Asthma (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 9 (16)
Lobar pneumonia (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4)
Pneumonia viral (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Bronchitis viral (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Parainfluenza virus infection (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Influenza (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Lupus pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cellulitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic sinusitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
H1N1 influenza (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Lung adenocarcinoma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Lung neoplasm malignant (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Metapneumovirus infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonia respiratory syncytial viral (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonia streptococcal (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory tract hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (4)
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Respiratory syncytial virus infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (5)
Acute sinusitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Lower respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonia bacterial (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonia haemophilus (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonia staphylococcal (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory syncytial virus test positive (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rhinovirus infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Squamous cell carcinoma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Tracheobronchitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tyvaso (N=666) | Control (N=667)
Cough (Respiratory, thoracic and mediastinal disorders) | 122 (155) | 106 (119)
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 99 (129) | 115 (158)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 89 (117) | 80 (109)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 57 (75) | 56 (73)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 55 (63) | 66 (85)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 55 (62) | 54 (70)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 50 (62) | 61 (81)
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 44 (55) | 48 (63)
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 41 (52) | 63 (73)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 39 (43) | 12 (13)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 37 (43) | 30 (32)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 26 (31) | 37 (37)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the United Therapeutics publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.